CLINICAL TRIAL: NCT04176913
Title: A Study Evaluating the Safety, Tolerability, and Pharmacokinetics of LUCAR-20S in Patients With Relapsed/Refractory Diffuse Large B-Cell, Follicular, Mantle Cell or Small Lymphocytic Lymphoma
Brief Title: Study of LUCAR-20S in Patients With R/R NHL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Both the sponsors and collaborator are considering terminating the study
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Legend Biotechnology Co.,Ltd.; The First Affiliated Hospital of USTC west district; Beijing Boren Hospital (Unknown)
Responsible Party: Principal Investigator, WEI XU, Chief Physician of hematology department, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM2L201904; BM2L201904 (Registry Identifier: BM2L201904); NCT04994587 (obsolete NCT alias)
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD20 Allogeneic CAR-T Cell Therapy (Experimental): An open label, single arm Phase I study to evaluate the safety, tolerability, and pharmacokinetics of LUCAR-20S CAR-T cells in relapsed or refractory CD20+ diffuse large B-cell, follicular, mantle cell and small lymphocytic lymphoma.
  Interventions: Drug: LUCAR-20S CAR-T cells

INTERVENTIONS:
Drug: LUCAR-20S CAR-T cells — An Anti-CD20 Allogeneic CAR-T Cell Therapy in Patients with Relapsed/Refractory Diffuse Large B-Cell, Follicular, Mantle Cell or Small Lymphocytic Lymphoma

SUMMARY:
An open label, single arm Phase I study to evaluate the safety, tolerability, and pharmacokinetics of LUCAR-20S CAR-T cells in relapsed or refractory CD20+ diffuse large B-cell, follicular, mantle cell and small lymphocytic lymphoma.

DETAILED DESCRIPTION:
This study is an open, dose escalation/dose regimen finding study to assess the safety and pharmacokinetics of donor-derived CD20-directed CAR-T cells administered with lymphodepletion, and to obtain the preliminary efficacy results in subjects who have been diagnosed with relapsed or refractory CD20 positive diffuse large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma or small lymphocytic lymphoma. The allo-CAR-T cells will be infused in single-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF)
2. Age 18 Years to 75 Years
3. Pathological diagnosis of refractory/relapsed CD20+ non-Hodgkin's lymphoma (one of the following):

   1. Diffuse large B-cell lymphoma (DLBCL)
   2. Follicular lymphoma (FL)
   3. Mantle cell lymphoma (MCL)
   4. Small lymphocytic lymphoma (SLL)
4. Measurable disease as defined by 2014 Lugano criteria at Screening
5. Refractory/relapsed disease after standard-of- care treatment as following (Undergone at least 2 complete cycle of therapy for each line, unless PD been documented as the best response to the regimen) and not eligible or appropriate for HSCT (Auto/allo). Subject must have documented evidence of progressive disease on or within 12 months of their last regimen.

   1. DLBCL: Refractory/relapsed after at least 1 prior line of therapy, must have been treated with anti-CD20 monoclonal antibody
   2. FL: Refractory/relapsed after at least 2 prior lines of therapy, must have been treated with anti-CD20 monoclonal antibody
   3. MCL: Refractory/relapsed after at least 2 prior lines of therapy
   4. SLL: Refractory/relapsed after at least 2 prior lines of therapy
6. Laboratory criteria at Screening

   ① Blood routine: NE≥1.0×109/L；HGB≥8g/dL；PLT≥50×109/L

   ② Blood biochemical parameters:
   1. Total bilirubin ≤ 1.5 times of the normal upper limit (ULN)
   2. Aspartate and alanine aminotransferases (AST, ALT) ≤ 3 times ULN (in the presence of liver metastasis, ULN 5 times)
   3. Estimated glomerular filtration rate (eGFR) > 60mL/min
7. Life expectancy > 12 weeks
8. Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 or 1

Exclusion Criteria:

1. Any malignancy besides the NHL categories under study, exceptions include

   1. Any other malignancy curatively treated and disease-free for at least 2 years prior to enrollment
   2. History of non-melanoma skin cancer with sufficient treatment and currently no evidence of recurrence
2. Prior treatment with an allogeneic stem cell transplant
3. Prior treatment with genetic therapy
4. Prior treatment with chimeric antigen receptor T (cells) CAR-T therapy directed at CD20 target
5. Those who are positive for any index of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), and human immunodeficiency virus antibody (HIV-Ab)
6. Prior antitumor therapy with insufficient washout period

   1. Targeted therapy, epigenetic therapy, experimental drug therapy or experimental invasive treatment with medical apparatus and instruments 14 days or five half-lives, whichever is shorter before lymphodepletion
   2. Use of monoclonal antibodies 21 days prior to lymphodepletion
   3. Chemotherapy within 14 days prior to lymphodepletion
   4. Radiotherapy within 14 days prior to lymphodepletion
   5. Participated in other clinical trials within 30 days prior to lymphodepletion
7. With central nervous system involvement
8. Women in pregnancy or lactation
9. Being fertile and unable to use effective conception during treatment and 100 days after CAR-T infusion
10. Active autoimmune disease or history of autoimmune disease within 3 years
11. With obvious hemorrhagic tendency such as gastrointestinal hemorrhage, coagulation disorders and hypersplenism
12. The following cardiac conditions

    1. New York Heart Association (NYHA) stage III or IV congestive heart failure
    2. Left ventricular ejection fraction (LVEF) less than (<)45%
    3. Uncontrolled cardiac arrhythmia post-medication
    4. With a history of myocardial infraction or unstable angina pectoris within the past 6 months
    5. Constrictive pericarditis
    6. Cardiomyopathy
13. Pulse oximetry of <96% on room air
14. Active or uncontrolled infection requiring parenteral antibiotics, or any evidence of severe active viral/bacterial infection or uncontrolled systemic fungal infection
15. Uncontrolled diabetes mellitus, defined as fast serum glucose > 1.5 times ULN
16. Concurrent use of corticosteroids or other immunosuppressant medications for chronic disease
17. Concurrent use of hematopoietic growth factor
18. Stroke or seizure within 6 months of signing ICF
19. Have received any live, attenuated vaccine within 4 weeks prior to lymphodepletion
20. Have underwent major surgical operation within 2 weeks prior to lymphodepletion, or anticipate to undergo a major surgical operation during the study process or within 2 weeks posterior to study treatment(with the exception of anticipated local anesthesia surgery)
21. Known life threatening allergies, hypersensitivity, or intolerance to LUCAR-20S CAR-T cells or its excipients, including dimethyl sulfoxide (DMSO)
22. Presence of any condition that, in the opinion of the investigator, would prohibit the patient from undergoing treatment under this protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 30 days post infusion
  DLT assessed by NCI-CTCAE 5.0
Adverse events | 90 days post infusion
  Incidence and severity of adverse events as assessed by NCI-CTCAE 5.0
Concentration of Pharmacokinetics in blood | through study completion, 2 years after infusion of the last subject
  PK CAR positive T cells in peripheral blood, PK CAR transgene levels in peripheral blood
Concentration of Pharmacokinetics in bone marrow | through study completion, 2 years after infusion of the last subject
  PK CAR positive T cells in bone marrow, PK CAR transgene levels in bone marrow

SECONDARY OUTCOMES:
Recommended Phase II dose (RP2D) | 30 days post infusion
  RP2D established through ATD+BOIN design and the DLTs occurring following CAR T-cell infusion
Overall response rate (ORR) after administration | 3 months post infusion
  Antitumor efficacy by 2014 Lugano criteria
Time to Response (TTR) after administration | 3 months post infusion
  Antitumor efficacy by 2014 Lugano criteria
Duration of remission (DOR) after administration | through study completion, 2 years after infusion of the last subject
  Antitumor efficacy by 2014 Lugano criteria
Progress Free Survival (PFS) after administration | through study completion, 2 years after infusion of the last subject
  Antitumor efficacy by 2014 Lugano criteria
Overall Survival (OS) after administration | through study completion, 2 years after infusion of the last subject
  Antitumor efficacy by 2014 Lugano criteria

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, PhD& MD, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital); Kaiyang Ding, PhD& MD, Principal Investigator — Anhui Provincial Cancer Hospital; Kai Hu, PhD& MD, Principal Investigator — Beijing Boren Hospital
Locations (3):
- China (3):
  - Oncology Department，The First Affiliated Hospital of USTC west district, Hefei, Anhui
  - Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu
  - Hematological Department，Beijing Boren Hospital, Beijing